CLINICAL TRIAL: NCT03043040
Title: Prevention of Suicidal Behaviour in High Risk Patients With Telemedicine Techniques
Brief Title: Prevention of Suicidal Behaviour With Telemedicine Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osakidetza (Other)
Collaborators: Eusko Jaurlaritza (Unknown)
Responsible Party: Principal Investigator, Andrea Gabilondo, Principal Investigator, Osakidetza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017AG01
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Suicide, Attempted
Keywords: suicide, attempted; prevention; telemedicine
MeSH Terms: conditions — Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a non-randomized non-blinded multicenter intervention study with control group. Patients from hospital A and B are included in the intervention group. Patients from hospital C are included in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone follow up (Experimental): Patients discharged from hospital A and B after a suicide attempt receive a protocolized telephone follow which is added to their usual treatment (TAU). Calls are made by nurses at weeks 1,2,4,12 and 24 after the index suicide attempt.
  TAU: Includes whatever treatment the doctor decides to offer to that patient (psychopharmacology, psychotherapy etc).
  Interventions: Behavioral: Telephone follow up; Behavioral: Treatment as usual
- Control (Active Comparator): Patients discharged from hospital C after a suicide attempt receive treatment as usual (whatever treatment the doctor decides to offer to that patient: psychopharmacology, psychotherapy etc).
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Telephone follow up — Already described in previous page
  Arms: Telephone follow up
Behavioral: Treatment as usual — Already described in previous page

SUMMARY:
This is a multicenter controlled intervention study that aims to assess the efficacy of a telephone follow-up program for the prevention of suicidal behavior in adults discharged from general hospitals after a suicide attempt.

The hypothesis is that the implementation of this program is associated with reduced rates of suicide reattempts in these patients and also with delayed reattempts in them.

DETAILED DESCRIPTION:
Justification: Suicide is a global public health concern and is the leading cause of avoidable death in the Basque Country (Spain). The use of telemedicine techniques applied to high risk patients has shown to be useful in the prevention of suicide and suicidal behavior.

Objectives: To assess the efficacy of a telephone follow-up program for the prevention of suicidal behavior in patients who recently attempted suicide.

Design: This is a multicenter, prospective intervention study, non-randomized and with control group.

Method: A sample of adults discharged from 2 general hospitals after a suicide attempt are enrolled in a telephone follow-up program which is added to their usual treatment (TAU). The program consists of 5 short calls made by nurses during 6 months. The calls are intended to: 1) Assess the risk of suicide in that moment, 2) Improve patient's adherence to treatments, and 3) Provide general psychoeducation guidelines. The control group is composed of patients discharged from a third general hospital after a suicide attempt. These receive TAU but are not enrolled in the telephone follow-up.

Evaluation: All patients are followed during 12 months. Main outcome measures include the percentage of patients that make a second attempt and the average time to reattempt.

Patients sign and informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients discharged from a General Hospital after a suicide attempt and who live in the same health sector as the hospital.
* The suicide attempt must have been made within 24 hours prior to the appointment in the Emergency Service.

Exclusion Criteria:

* Patient with severe cognitive difficulties and in general any self-injury in which the patient does not understand the meaning or potential consequences of such behavior.
* Patients in which a regular telephone contact is not possible.
* Patients in which the psychiatrist who evaluates the case deems inappropriate their inclusion.
* Patients who remain hospitalized 6 months after the attempt.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants in each group that make a second attempt | 0-12 months
  (Included in the title)

SECONDARY OUTCOMES:
Average number of days from the first attempt to the second, in each group | 0-12 months
  (Included in the title)
Mean number of reattempts in each group | 0-12 months
  (Included in the title)
Percentage of participants in each group requiring hospitalization after the suicide attempt | 0-12 months
  (Included in the title)

IPD SHARING:
Plan to Share IPD: No